CLINICAL TRIAL: NCT04778748
Title: Evaluating an Under-mattress Sleep Monitor Compared to a Peripheral Arterial Tonometry Home Sleep Apnea Test Device in the Diagnosis of Obstructive Sleep Apnea
Brief Title: Evaluating an Under-mattress Sleep Monitor Compared to a Peripheral Arterial Tonometry Device in the Diagnosis of Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Withings (Industry)
Responsible Party: Principal Investigator, Timothy Morgenthaler, Principal Investigator, Mayo Clinic
Other Study IDs: 20-010024
Record Dates: First submitted 2021-01-29; First posted 2021-03-03 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstructive Sleep Apnea: Participants will be provided with a Withings sleep monitor and instructed to begin using it. Effective data collection via the Withings unit should be confirmed for at least 7 consecutive nights, and the WatchPAT device will be used during one of those same 7 nights.
  Interventions: Diagnostic Test: Under-mattress sleep monitor

INTERVENTIONS:
Diagnostic Test: Under-mattress sleep monitor — Under-mattress sleep monitor for patients with a confirmed diagnosis of Obstructive Sleep Apnea.

SUMMARY:
A device has been developed which is placed under the mattress, thereby escaping contact with patient, which enables monitoring of sleep activity and has been shown in some studies to provide an estimate of the frequency of sleep disordered breathing. If the estimates of sleep disordered breathing from this new device are medically equivalent to current excepted home sleep apnea test devices within clinically important ranges of sleep disordered breathing, it may have several benefits. This study is designed to help answer several important clinical questions, namely, is the new device clinically equivalent to an established HSAT device for patients who have at least moderately severe OSA, and what is the effect of multiple nights on classification of severity and presence of OSA.

DETAILED DESCRIPTION:
The design will be a prospective test of two diagnostic testing strategies. The tests will take place in the same patient concurrently, so the patient's results from one test will serve as the comparator with the other test device. No randomization or blinding is needed.

Patients will be recruited from the Mayo Clinic Center for Sleep Medicine (and another sleep center with enriched racial variety). Consecutive patients in whom the clinician has ordered a WatchPAT™ will be potential candidates for an opportunity to participate in the study. Patients will be made aware of the trial by invitation from members of the healthcare team. Interested patients will be evaluated according to the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

Clinician suspects of having OSA due to presence of any:

* STOP-BANG ≥ 3,
* overnight oximetry with ODI ≥ 5,
* STOP-BANG≥ 2 and one or more of: disrupted sleep, cognitive complaints, paroxysmal or prior atrial-fibrillation (now in NSR), stroke, TIA
* Has a smartphone capable of running both Withings and Itamar's app
* Stable sleeping quarters and schedule (i.e., no overnight shifts) for at least 7 days
* Domicile has capable wireless internet service

Exclusion Criteria:

* Uses short-acting nitrates within 3 hours of the study
* Has a permanent pacemaker
* Atrial fibrillation or sustained supraventricular arrhythmias
* Known congestive heart failure Class ≥ 1, or known LVEF< 45%
* Sustained hypoxemia or hypoventilation (results of RA daytime ABG show SaO2<90% or PaCO2>45 mmHg, or overnight oximetry shows mean SaO2<90%.)
* Advanced pulmonary disease (COPD GOLD stage ≥ II , pulmonary fibrosis with GAP ≥ 1 or significant dyspnea on exertion

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of OSA
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
The apnea hypopnea index (AHI) | 12 months
  The apnea hypopnea index (AHI) provided by one-night of testing with the WatchPAT™ is equivalent to the AHI provided by the mean of 7 nights use of the Withings™ sleep monitor. The equivalence margin will be an AHI≤5/hr.

SECONDARY OUTCOMES:
Sensitivity | 12 months
  The Withings sleep monitor will have a sensitivity ≥ 0.825 to identify patients with moderate to severe OSA as assessed by a WatchPAT AHI≥15.

OTHER OUTCOMES:
Positive likelihood ratio | 12 months
  The Withings sleep monitor will have a likelihood ratio ≥ 5 to identify patients with moderate to severe OSA as assessed by a WatchPAT AHI≥15

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Morgenthaler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linz D, Baumert M, Desteghe L, Kadhim K, Vernooy K, Kalman JM, Dobrev D, Arzt M, Sastry M, Crijns HJGM, Schotten U, Cowie MR, McEvoy RD, Heidbuchel H, Hendriks J, Sanders P, Lau DH. Nightly sleep apnea severity in patients with atrial fibrillation: Potential applications of long-term sleep apnea monitoring. Int J Cardiol Heart Vasc. 2019 Oct 18;24:100424. doi: 10.1016/j.ijcha.2019.100424. eCollection 2019 Sep. PMID 31763438
- [Background] Sadek I, Biswas J, Abdulrazak B. Ballistocardiogram signal processing: a review. Health Inf Sci Syst. 2019 May 16;7(1):10. doi: 10.1007/s13755-019-0071-7. eCollection 2019 Dec. PMID 31114676
- [Background] Walsh L, McLoone S, Ronda J, Duffy JF, Czeisler CA. Noncontact Pressure-Based Sleep/Wake Discrimination. IEEE Trans Biomed Eng. 2017 Aug;64(8):1750-1760. doi: 10.1109/TBME.2016.2621066. Epub 2016 Oct 25. PMID 27845651
- [Derived] Jagielski JT, Bibi N, Gay PC, Junna MR, Carvalho DZ, Williams JA, Morgenthaler TI. Evaluating an under-mattress sleep monitor compared to a peripheral arterial tonometry home sleep apnea test device in the diagnosis of obstructive sleep apnea. Sleep Breath. 2023 Aug;27(4):1433-1441. doi: 10.1007/s11325-022-02751-7. Epub 2022 Nov 28. PMID 36441446
- See also: Patent — https://data.epo.org/publication-server/rest/v1.2/patents/EP3763290NWA1/document.html
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials